CLINICAL TRIAL: NCT00822887
Title: A Phase I Dose Escalation Study of Vandetanib (ZACTIMA, ZD6474) With Hypofractionated Stereotactic Radiotherapy in Patients With Recurrent Malignant Gliomas
Brief Title: Dose Escalation Study of Vandetanib With Hypofractionated Stereotactic Radiotherapy in Recurrent Malignant Gliomas
Acronym: IRUSZACT0073
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0870.cc; NCT00721292 (obsolete NCT alias)
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Gliomas
Keywords: malignant; gliomas
MeSH Terms: conditions — Glioma | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib (Experimental): Dose level 1:100 mg qd, 2:200 mg qd, 3:300 mg qd. Fractionated Stereotactic Radiotherapy: all patients will receive 36 Gy of radiation in three fractions, given in three consecutive days.
  Interventions: Drug: Vandetanib; Radiation: Fractionated Stereotactic Radiotherapy

INTERVENTIONS:
Drug: Vandetanib — Dose level 1:100 mg qd Dose level 2:200 mg qd Dose level 3:300 mg qd
  Other Names: ZD6474, Zactima
Radiation: Fractionated Stereotactic Radiotherapy — All patients will receive 36 Gy of radiation in three fractions, given in three consecutive days.

SUMMARY:
The purpose of the study is to find out the highest dose of vandetanib that can be safely given with repeat radiation therapy.

This study drug has been designed to block certain chemical pathways that stimulate tumor to grow. The study drug has been shown to slow the growth of a number of types of cancers.

This will be a dose escalation study. A dose escalation study means that successive groups of patients will receive higher doses of the study drug. There are three dose levels. The dose of the study drug received will depend on the stage the study has reached at the time a patient decides to participate.

In addition to taking the study drug patients will also receive radiation therapy to the brain tumor for 3 days.

Hypothesis The objective of this study is to determine the maximally tolerated dose (MTD) of VANDETANIB given with 36 Gy hypofractionated stereotactic radiotherapy. The MTD will be dose of VANDETANIB at which no patients develop acute grade 5 toxicity and less than 30% of patients develop acute (within 30 days of radiation therapy) or delayed (at least 30 days after radiation completed) dose limiting toxicities.

DETAILED DESCRIPTION:
Screening Prior to receiving any treatment, tests will be performed to determine overall medical condition. This will include blood tests, questions about medical history, and physical and neurological exams.

MRI scan of the brain, electrocardiogram (ECG) and chest X-ray will be performed as baseline studies if they have not been performed in the last 28 days.

Women of child-bearing potential will also have a serum pregnancy test within 2 days before taking the study drug.

During treatment If all of the study criteria are met and subject is enrolled in the study, you will start taking the study drug at least 7 days before radiation therapy. You will take the study drug once a day by mouth. You should take the study drug at about the same time each day. If you forget to take a dose, take the missed dose as soon as you remember, as long as it is at least 12 hours before the next dose is due. If it is less than 12 hours until the next dose, do not take the dose you have missed. If you throw up within 30 minutes after you take the study drug, you should take another dose, and use medicine to stop or relieve your vomiting per your doctor's instruction. You will continue to take the study drug for a total duration of one year. The study will be stopped if your disease progresses or there is excessive toxicity. Your participation in the study will be for one year. However, we will continue to follow your disease status, general health and possible treatment-related side effects after one year and for as long as possible.

This is a Phase I study. These types of studies usually include a small number of subjects and are often called dose-escalation studies. Subjects in the first dose group will be receiving a small dose of the study drug. If no unacceptable side effects are observed in these subjects, the next group of subjects will receive the next higher dose of study drug. The study drug doses planned are as follows:

Dose Level Drug dose Level 1 100 mg once a day Level 2 200 mg once a day Level 3 300 mg once a day

You will be assigned to one of three levels depending on when you enter the study.

You will also receive radiation therapy. The radiation dose is the same for all patients. Radiation therapy will begin at least 7 days after you begin taking the study drug. The radiation therapy will be once a day for 3 consecutive days. A special plastic mask will be made for you and used to hold your head still during each radiation treatment.

Tests and procedures will be performed throughout your treatment to determine how your cancer is responding and to monitor you for safety purposes. The tests and procedures will be scheduled for you. The following tests and procedures will be performed:

* Physical examination, neurological examination, and ECG, right before, and in the first, second, fourth, eighth and twelfth week of drug treatment; then once every three months.
* Brain MRI and quality of life questionnaires at one month and three month after radiation therapy, then once every three months.
* Chest X-ray as your doctor determines.

Follow-up You will also have follow-up visits with your doctor once a month for the first 6 months, then once every three months. You may also see your doctor anytime as needed.

Duration You will be on this study for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically confirmed malignant gliomas that recurred after surgical resection and conventional radiation therapy
* Tumor is not located in the eloquent part of the brain and not touching the brainstem, optic chiasm or optic nerve so that these critical structures will not receive full dose of re-irradiation
* Recurrent tumor is not surgically resectable or patient is not medically operable
* Age > 18 years.
* Radiographical evidence of local recurrence on brain MRI, with or without histopathological confirmation.
* Estimated survival of at least 3 months
* Zubrod Performance Scale of 0-2
* Hgb greater than 10 gm/dl, absolute neutrophil count greater than 1500/ul, platelets greater than 100,000/ul, blood urea nitrogen (BUN) less than 25 mg/dl, Bilirubin less than 2.0 mg/dl, serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) less than 2 x normal range
* Less than or equal to 3 recurrent tumors, and combined largest diameter of all tumors less than or equal to 6 cm
* Single recurrent tumor less than or equal to 6 cm in the largest diameter

Exclusion Criteria:

* Prior therapy with any anti-Epidermal growth factor receptor(EGFR) and/or anti-VEGFR therapies
* Recurrent tumor greater than 6 cm in the largest diameter
* Recurrent tumor located in the brainstem.
* Prior radiation therapy to the brain within 2 months.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition (such as severe cognitive impairment)
* pregnant and breast-feeding women will be excluded
* Treated on any other clinical protocols or with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)
* Clinically significant cardiac event
* History of arrhythmia. Atrial fibrillation, controlled on medication is not excluded.
* Previous history of corrected electrocardiogram QT interval (QTc)prolongation as a result from other medication that required discontinuation of that medication.
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block QTc with Bazett's correction that is unmeasurable, or 480 msec on screening ECG. If a patient has QTc 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than 480 msec in order for the patient to be eligible for the study.
* Concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce cytochrome P450 3A4 (CYP3A4) function Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
* Active diarrhea that may affect the ability of the patient to absorb the VANDETANIB.
* Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy
* Clinical and/or radiographic evidence of bleeding in the recurrent brain tumor.
* Patients currently on enzyme inducing anticonvulsants. However, patients are eligible if the enzyme inducing anticonvulsants can be discontinued or switched to non- enzyme inducing anticonvulsants one week before study entry. Non-enzyme inducing anticonvulsants cannot be those which may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
* Laboratory results:

  * Serum bilirubin greater than 1.5 x the upper limit of reference range (ULRR)
  * Serum creatinine greater than 1.5 x ULRR or creatinine clearance less than 50 mL/minute (calculated by Cockcroft-Gault formula)
  * Potassium, less than 4.0 mmol/L despite supplementation; serum calcium (ionized or adjusted for albumin,) or magnesium out of normal range despite supplementation
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 X ULRR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of acute and delayed ≥ grade 3 Central nervous system (CNS) toxicity by Common Terminology Criteria (CTC) v.3. | 12 months.

SECONDARY OUTCOMES:
Incidence of acute and delayed ≥ grade 3 non-CNS toxicity | 12 months.
Progression-free survival at 6 months | 12 months.
Overall survival | 12 months.
Objective response rate | 12 months.
Quality of survival | 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Changhu Chen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Science Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Fields EC, Damek D, Gaspar LE, Liu AK, Kavanagh BD, Waziri A, Lillehei K, Chen C. Phase I dose escalation trial of vandetanib with fractionated radiosurgery in patients with recurrent malignant gliomas. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):51-7. doi: 10.1016/j.ijrobp.2010.09.008. Epub 2010 Oct 29. PMID 21035955